CLINICAL TRIAL: NCT05959720
Title: Adult Acute Lymphoblastic Leukemia Treated With Pediatric Regimen in Brazil - a Prospective Collaborative Study
Brief Title: Adult Acute Lymphoblastic Leukemia Treated With Pediatric Regimen in Brazil
Acronym: BRALLA
Status: Recruiting | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Wellington Fernandes, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Other Study IDs: 3011/22
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoid Leukemia; Minimal Residual Disease; Gene Abnormality; Chemotherapeutic Toxicity
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — Prednisone; Vincristine; Daunorubicin; pegaspargase; Cyclophosphamide; Cytarabine; Mercaptopurine; Methotrexate; Doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — All bone marrow or peripheral blood samples from diagnosis are going to be stored in a registered biobank. From bone marrow, DNA, RNA (Trizol) and mononuclear cryopreserved cells are going to be stored after Ficoll separated centrifugation. From peripheral blood, only DNA/RNA from buffy coat.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Eligible patients: All patients deemed eligible to intensive protocol of treatment are going to be included as sole group. There is no intervention or control group in this trial.
  Interventions: Drug: Prednisone; Drug: Vincristin; Drug: Daunorubicin; Drug: Peg-asparaginase; Drug: Intrathecal Suspension; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Doxorubicin

INTERVENTIONS:
Drug: Prednisone — 60 mg/m2 D1 to D21
Drug: Vincristin — 1.5 mg/m2 D1, D8, D15 and D22
Drug: Daunorubicin — 40 mg/m2 D1, D8, D15 and D22
Drug: Peg-asparaginase — 2000 UI/m2 D12 and D26
Drug: Intrathecal Suspension — MTX 12 mg, Dexamethasone 2 mg, Cytarabine 60 mg D1, D8, D15, D22, D29
Drug: Cyclophosphamide — 1000 mg/m2 D36 and D64
Drug: Cytarabine — 75 mg/m2 D36 to D39, D43 to D46, D50 to D53 and D57 to D60
Drug: Mercaptopurine — 30 mg/m2 D36 to D63 and D1 to D56 of consolidation
Drug: Methotrexate — 3.000 mg/m2 D8, D22, D36 and D50
Drug: Doxorubicin — 30 mg/m2 D1 and D22

SUMMARY:
In this project, the investigators intend to start a prospective registry for patients with newly diagnosed Philadelphia-negative ALL from 16 years old and above in participating centers, provided that all patients will be treated with the same regimen (a pediatric regimen BFM-based incorporating peg-asparaginase). All diagnostic/follow-up (after induction and consolidation blocks) samples will be centrally biobanked at Instituto do Cancer do Estado de Sao Paulo. The main goal of this study is to examine whether the implementation of a pediatric protocol under a prospective registry can increase event-free survival (EFS) and overall survival (OS) of newly diagnosed patients in the participating centers.

DETAILED DESCRIPTION:
Notably, pediatric regimens for adult acute lymphoblastic leukemia (ALL) have resulted in better long-term outcomes, especially in the Philadelphia-negative counterpart. These regimens are essentially based on higher cumulative doses of asparaginase and the use of less myelotoxic agents, applying allogeneic transplantation only for high-risk ALL subsets. Recent metanalysis encompassing 27 clinical trials demonstrated an improved prognosis when these regimens are adopted. In adults, incorporation of these regimens has been hampered by a perception of higher toxicity and a more complex design, especially with asparaginase. Remarkably, this drug might bring side effects not usually seen with other cancer drugs, such as thrombosis, liver, and pancreatic toxicities. In addition, the incorporation of minimal residual disease (MRD) monitoring throughout the treatment protocol in a scheduled and standardized manner is considered paramount in the contemporary ALL treatment. Treating adult patients with acute leukemia under prospective studies allows accurate data collection and positively impacts the disease prognosis, creating a cooperative scientific environment. In Brazil, few data are available on the clinical- laboratory characteristics of ALL in adults and their outcomes under a standardized treatment protocol. Few single-center reports point to a worse overall survival rate when compared to developed countries. There is great heterogeneity across the centers regarding the treatment regimens and genetic/MRD assessment. In this project, the investigators intend to start a prospective registry for patients with newly diagnosed Philadelphia-negative ALL from 16 years old and above in participating centers, provided that all patients will be treated with the same regimen (a pediatric regimen BFM-based incorporating peg-asparaginase). All diagnostic/follow-up (after induction and consolidation blocks) samples will be centrally biobanked at Instituto do Cancer do Estado de Sao Paulo. At the diagnosis, a genetic characterization encompassing conventional karyotype, fluorescent in-situ hybridization (FISH), and molecular biology in our central laboratory will be performed to classify the cases. Genomic classification will include identifying Philadelphia- like B-cell ALL cases, a recent group of cases with worse prognosis, whose incidence seems higher in Hispanics. In Brazil, there is no study addressing this incidence and, more importantly, evaluating its impact on outcomes under a standardized treatment protocol. MRD analysis will also be centralized to standardize and validate our flow cytometry panel in a homogeneous cohort. Additionally, the investigators plan to assess baseline factors predictive of survival and relapse and those related to major toxicities such as infections, liver toxicity, and thrombosis.

ELIGIBILITY:
Inclusion Criteria: Patients between 16 and 50 years-old with newly diagnosed ALL, negative for Philadelphia chromosome not previously treated (except for hydroxyurea, corticosteroids, or intrathecal chemotherapy) with 20% or more lymphoblasts in bone marrow or peripheral blood.

Exclusion Criteria:

* Burkitt leukemia
* Prior myeloproliferative disease
* Philadelphia chromosome positivity through whichever methodology (RT-PCR, FISH, or conventional karyotype)
* ECOG>2 (appendix 3)
* Total bilirubin>2x upper limit of normal (ULN)
* Transaminases>5x ULN
* Creatinine>2,5 mg/dl
* Positive serology for HIV or HTLV
* Heart failure NYHA Class III or IV (appendix 4)
* Severe psychiatric disorder which prevents adequate compliance
* Prior treatment with intravenous chemotherapy
* Refusal to participate in the study
* Down syndrome

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients from 16 years and above newly diagnosed with Philadelphia-negative ALL and after the signature of informed consent form (ICF). Patients between 16 and 17 years-old will sign a child assent along with a parental consent form. ICF application might be performed even under ALL suspicion only, given the need for sample collection before any therapy, ideally.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 4 years
  cumulative proportion of patients alive (considering the time between the date of diagnosis and death or last follow-up)

SECONDARY OUTCOMES:
Event-free survival (EFS) | 4 years
  time between enrollment in the study and the occurrence of any event: refractoriness after the first two cycles of induction, death or relapse.
Early death rate | 60 days
  proportion of patients who died before the first bone marrow evaluation of response (after induction I)
Complete response rate | 60 days
  proportion of patients with bone marrow aspirate with less than 5% blasts and evidence of normal hematopoiesis; CSF without blasts and recovery of peripheral blood (neutrophils≥ 1,000/μL and platelets≥100,000/μL), without the need for transfusion
Cumulative incidence of relapse | 4 years
  rate of disease relapse after CR calculated considering death as a competing event.
HSCT rate | 2 years
  proportion of patients eligible for the protocol who were able to perform the procedure in their first CR

CONTACTS AND LOCATIONS:
Overall Officials: Wellington F Silva, MD PhD, Principal Investigator — Instituto do Cancer do Estado de São Paulo; Eduardo M Rego, MD PhD, Study Chair — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Silva WF, Amano MT, Perruso LL, Cordeiro MG, Kishimoto RK, de Medeiros Leal A, Nardinelli L, Bendit I, Velloso ED, Rego EM, Rocha V. Adult acute lymphoblastic leukemia in a resource-constrained setting: outcomes after expansion of genetic evaluation. Hematology. 2022 Dec;27(1):396-403. doi: 10.1080/16078454.2022.2052602. PMID 35344469